CLINICAL TRIAL: NCT03736512
Title: Prospective Registry of Outcomes With the GreenLight™ Laser System
Brief Title: China Greenlight Registry Study (Post-market)
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: U0597
Record Dates: First submitted 2017-09-04; First posted 2018-11-09 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Benign Prostatic Hyperplasia (BPH)
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Device: GreenLight XPS™ 532 nm Laser System with MoXy™ laser fiber — observational registry

SUMMARY:
The duration of the study is expected to take approximately 3 years, which includes a recruitment period of approximately 12-months and 2 years (24-months) to complete procedure and follow-up visits.

DETAILED DESCRIPTION:
The study follow-up duration from the primary study procedure is 5 years.

* Baseline
* Study Procedure
* 4-week
* 6-month
* 12-month
* 24-month (End of Study) The study will be considered complete after all subjects have completed the 24-month follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent and agrees to attend all study visits
* Subject has a diagnosis of lower urinary tract symptoms due to benign prostatic enlargement causing bladder outlet obstruction
* Subject is able to complete self-administered questionnaires
* Clinical investigator has documented in the subject's medical record that in his/her judgment the subject is a surgical candidate for the PVP procedure
* Subject is ≥ 40 years of age
* Subject has an IPSS score greater than or equal to 12 measured at the baseline visit
* Subject has medical record documentation of a maximum urinary flow rate (Qmax) less than or equal to 15ml/s and sample is greater than or equal to 150ml (If uroflow testing documentation is available within 90 days prior to the informed consent date, and the sample is greater than or equal to 150ml, and the Qmax is less than or equal to 15ml/s it may be used for the inclusion/exclusion criteria)
* Subject has medical record documentation of a prostate volume of greater than or equal to 30 grams by transrectal ultrasound (TRUS))

Exclusion Criteria:

* Subject has a life expectancy of less than 2 years
* Subject is classified as American Society of Anesthesiologists (ASA) V
* Subject is currently enrolled in, or plans to enroll in, any concurrent drug or device study unless preapproved by the sponsor
* Subject has an active infection that would preclude operation within 14 days of the study procedure (e.g., urinary tract infection or prostatitis)
* Subject has a diagnosis of, or has received treatment for, chronic prostatitis or chronic pelvic pain syndrome (e.g., non-bacterial chronic prostatitis)
* Subject has a neurogenic bladder or other neurological disorder that would impact bladder function (e.g., multiple sclerosis, Parkinson's disease, spinal cord injuries)
* Subject has a diagnosis of polyneuropathy (e.g., diabetic)
* Subject has diagnosis of stress urinary incontinence that requires treatment or daily pad/device use
* Subject has a diagnosis of prostate cancer or suspected prostate cancer based on PSA results and meeting the following:

PSA level of 4 - 10 with an abnormal DRE (if biopsy collected must be positive); PSA level greater than 10 with a positive biopsy

* Subject has a history of CIS, TaGIII or any T1 stage bladder cancer
* Subject has damage to external urinary sphincter
* Subject has had an acute myocardial infarction, open heart surgery or cardiac arrest less than 180 days prior to the date of informed consent
* Subject is immunocompromised (e.g., organ transplant, leukemia)
* Subject currently or has a history of upper urinary tract stones
* Subject currently diagnosed with OAB and treated with medication If the subject does not carry a diagnosis but is suspected to have OAB, the investigator must use his/her discretion

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Men diagnosed with benign prostatic hyperplasia (BPH) for whom GreenLight Laser therapy is recommended by their physician and eligible for inclusion.
Study Population: Men diagnosed with benign prostatic hyperplasia (BPH) for whom GreenLight Laser therapy is recommended by their physician and eligible for inclusion.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-11-29 (Actual)

PRIMARY OUTCOMES:
The GreenLight XPS system provides durable relief of BPH symptoms in subjects. | 6-month follow up
  Changes of IPSS Scores in subjects treated with the GreenLight XPS Laser System at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jian Huang, Doctor, Principal Investigator — Sun Yat-sen Memorial Hosptital, Sun Yat-sen University
Locations (1):
- Sun Yat-sen Memorial Hosptital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided